CLINICAL TRIAL: NCT00139100
Title: Evaluation of Antibacterial Soap for Treatment of Lymphedema and Elephantiasis in an Area Endemic for Lymphatic Filariasis
Brief Title: Evaluation of Antibacterial Soap for Treatment of Lymphedema in a Filariasis-Endemic Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Procter and Gamble (Industry); Ste. Croix Hospital, Leogane, Haiti (Unknown)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CDC-NCID-2822
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2005-08

CONDITIONS: Lymphedema; Cellulitis
MeSH Terms: conditions — Lymphedema; Cellulitis | interventions — Anti-Infective Agents; Soaps

INTERVENTIONS:
Drug: antimicrobial agent in soap

SUMMARY:
Introduction. Lymphatic filariasis is a devastating mosquito-transmitted parasitic disease that causes lymphedema or elephantiasis of the leg in 15 million persons, the majority of whom are women. In these persons, frequent bacterial infections ("acute attacks") of the legs adversely affect physical health, economic well-being, and quality of life. Prevention of bacterial infections through hygiene and skin care can result in significant improvements in lymphedema and patient well-being.

Methods. To determine the extent to which antibacterial soap can help reduce the incidence of acute bacterial infections of the lower limbs in persons with filarial lymphedema, 200 patients of the Ste. Croix Hospital lymphedema treatment clinic in Leogane, Haiti randomly assigned to receive either antibacterial (Safeguard) or placebo (Camay) soap and acute attacks monitored monthly for 12 months. Both groups received specific instructions on washing and skin care.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for participation include those who are currently enrolled in the lymphedema treatment program in Leogane who 1) have been trained in the techniques of self-care, 2) who live in a 10-km radius of the hospital, and 3) for whom we have adequate data on incidence of acute bacterial infections, risk factors for infection, and ability to comply with the treatment protocol (particularly hygiene).

-

Exclusion Criteria: Don't meet inclusion criteria.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2001-02; Study Completion 2002-03

PRIMARY OUTCOMES:
Incidence of bacterial "acute attacks", assessed monthly.
Reported or observed severity of these acute attacks.
Duration of acute attacks.

SECONDARY OUTCOMES:
Process measures
Number of bars of soap used per patient per month.
Demonstrated knowledge and ability to wash leg appropriately during home visits.
Reported patient satisfaction with soap.
Reported frequency of leg washing.

CONTACTS AND LOCATIONS:
Overall Officials: David G Addiss, MD, Principal Investigator — CDC/NCID/DPD
Locations (1):
- Hopital Ste. Croix, Léogâne, Haiti

REFERENCES:
- [Derived] Addiss DG, Michel MC, Michelus A, Radday J, Billhimer W, Louis-Charles J, Roberts JM, Kramp K, Dahl BA, Keswick B. Evaluation of antibacterial soap in the management of lymphoedema in Leogane, Haiti. Trans R Soc Trop Med Hyg. 2011 Jan;105(1):58-60. doi: 10.1016/j.trstmh.2010.08.011. Epub 2010 Sep 17. PMID 20850849